CLINICAL TRIAL: NCT02664740
Title: Comparison of the Efficacy of Standard Treatment Associated With Phage Therapy Versus Standard Treatment Plus Placebo for Diabetic Foot Ulcers Monoinfected by Staphylococcus Aureus: a Randomized, Multi-centre, Controlled, 2-parallel-group, Double-blind, Superiority Trial
Brief Title: Standard Treatment Associated With Phage Therapy Versus Placebo for Diabetic Foot Ulcers Infected by S. Aureus
Acronym: PhagoPied
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Collaborators: Phaxiam Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PHRC-N/2015/AS-01
Record Dates: First submitted 2016-01-19; First posted 2016-01-27 (Estimated); Last update posted 2022-02-03 (Actual); Status verified 2022-02

CONDITIONS: Diabetic Foot; Staphylococcal Infections
Keywords: Phage Therapy
MeSH Terms: conditions — Diabetic Foot; Staphylococcal Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Phage therapy (Experimental): Patients randomized to this arm will have phage therapy.
  Intervention: Topical anti-Staphylococcus bacteriophage therapy
  Interventions: Drug: Topical anti-Staphylococcus bacteriophage therapy
- Placebo (Placebo Comparator): Patients randomized to this arm will have placebo therapy anologous to that of the experimental arm.
  Intervention: Topical placebo corresponding to anti-Staphylococcus bacteriophage therapy
  Interventions: Drug: Topical placebo corresponding to anti-Staphylococcus bacteriophage therapy

INTERVENTIONS:
Drug: Topical anti-Staphylococcus bacteriophage therapy — Patients randomized to the experimental arm will receive sterile compress dressings impregnated with a phage solution of 10^7 PFU/ml on days 0, 7 and 14 (unless the wound is already healed, i.e. phage solutions are not applied to healed wounds).
  Arms: Phage therapy
Drug: Topical placebo corresponding to anti-Staphylococcus bacteriophage therapy — Patients randomized to the placebo arm will receive sterile compress dressings impregnated with a placebo solution on days 0, 7 and 14 (unless the wound is already healed, i.e. placebo solutions are not applied to healed wounds).
  Arms: Placebo

SUMMARY:
The primary objective of this study is to compare the efficacy of standard treatment associated with a topical anti-staphylococcal bacteriophage cocktail versus standard treatment plus placebo for diabetic foot ulcers monoinfected by methicillin-resistant or susceptible S. aureus (MRSA or MSSA) as measured by the relative reduction in wound surface area (%) at 12 weeks.

DETAILED DESCRIPTION:
The secondary objectives of this study are:

A. To compare the two study arms in terms of treatment safety and tolerance throughout the study.

B. To compare the two study arms in terms of further changes in wound healing at weeks 2, 4, 6, 8, 10, 12.

C. To describe the changes in the resistance and virulence of S. aureus (if present in the wound) from baseline to week 4, at modification of the first-line treatment or new antibiotic prescription (if any) and at week 12 if the wound is still not healed.

D. To describe in the two study arms the antibiotic resistance status of other bacteria isolated from wounds at week 4, at modification of the first-line treatment or new antibiotic prescription (if any) and at week 12 if the wound is still not healed.

E. To describe in the two study arms changes in wound microbiota from baseline to week 4, at modification of the first-line treatment or new antibiotic prescription (if any) and at week 12 if the wound is still not healed.

F. To describe the production of anti-phage antibodies during the topical treatment: baseline and week 4, at modification of the first-line treatment or new antibiotic prescription (if any), and at week 12.

G. Creation of a biobank for future ancillary studies (including, but not limited to, cytokine levels and cellular immune responses): days 0 and week 4, as well as week 12.

ELIGIBILITY:
Participant pre-inclusion criteria:

* The patient must have given his/her informed and signed consent
* The patient must be insured or beneficiary of a health insurance plan
* The patient is at least 18 years old
* The patient has type 1 or type 2 diabetes
* The patient is hospitalized/consulting in a participating centre
* The patient has a wound below the ankle that has be evolving for >2 weeks
* The target wound is classified as P (1 or 2), E (1-30 cm^2), D (2), I (2) and S (1 or 2) according to the PEDIS classification

Participant final inclusion criteria:

* The patient must have given his/her informed and signed consent
* The patient must be insured or beneficiary of a health insurance plan
* The patient is at least 18 years old
* The patient has type 1 or type 2 diabetes
* The patient is hospitalized/consulting in a participating centre
* The patient has a wound below the ankle that has be evolving for >2 weeks
* The target wound is classified as P (1 or 2), E (1-30 cm^2), D (2), I (2) and S (1 or 2) according to the PEDIS classification
* The patient's wound is mono-infected with Staphylococcus aureus (MRSA or MSSA)

Participant pre-exclusion criteria:

* The patient is participating in, or has participated in over the past three months, another trial
* The patient is participating in, or has participated in over the past three months, another study that may interfere with the results or conclusions of this study
* The patient is in an exclusion period determined by a previous study
* The patient is under judicial protection, or is an adult under guardianship
* It is impossible to correctly inform the patient
* The patient refuses to sign the consent
* The patient is pregnant, parturient or breastfeeding

Participant final exclusion criteria:

* The patient is participating in, or has participated in over the past three months, another trial
* The patient is participating in, or has participated in over the past three months, another study that may interfere with the results or conclusions of this study
* The patient is in an exclusion period determined by a previous study
* The patient is under judicial protection, or is an adult under guardianship
* It is impossible to correctly inform the patient
* The patient refuses to sign the consent
* The patient is pregnant, parturient or breastfeeding
* Patients who have received antibiotics within the 7 days preceding inclusion
* Patients with diabetic foot wounds associated with clinical or radiographic signs of arthritis or osteomyelitis*
* Patients with diabetic foot wounds associated with critical limb ischemia according to P = grade 3 in the PEDIS classification
* Patients whose wound is infected by a pathogen other than S. aureus (includes multi-infections) according to bacteriological sampling performed at the pre-inclusion visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-06-01 (Estimated); Primary Completion 2024-08 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
The relative reduction in wound surface area (%) | 12 weeks

SECONDARY OUTCOMES:
Immediate Safety | Day 0, 1 hour after application of experimental dressing
  The presence/absence of the following symptoms during each 1 hour observation periods following the application of each experimental wound dressing: local side effects (local rash onset or worsening of local inflammatory signs) and general symptoms (vital signs, fever, rash, arthralgia, gastro-intestinal symptoms...) will be performed.
Immediate Safety | Day 7, 1 hour after application of experimental dressing
  The presence/absence of the following symptoms during each 1 hour observation periods following the application of each experimental wound dressing: local side effects (local rash onset or worsening of local inflammatory signs) and general symptoms (vital signs, fever, rash, arthralgia, gastro-intestinal symptoms...) will be performed.
Immediate Safety | Day 14, 1 hour after application of experimental dressing
  The presence/absence of the following symptoms during each 1 hour observation periods following the application of each experimental wound dressing: local side effects (local rash onset or worsening of local inflammatory signs) and general symptoms (vital signs, fever, rash, arthralgia, gastro-intestinal symptoms...) will be performed.
The number of MedDRA coded Adverse Events per patient | throughout the study; 12 weeks
The presence/absence of abnormal laboratory results | throughout the study; 12 weeks
Wound surface area | 2 weeks
Wound surface area | 4 weeks
Wound surface area | 6 weeks
Wound surface area | 8 weeks
Wound surface area | 10 weeks
Wound surface area | 12 weeks
Wound depth | 2 weeks
Wound depth | 4 weeks
Wound depth | 6 weeks
Wound depth | 8 weeks
Wound depth | 10 weeks
Wound depth | 12 weeks
Time to healing | censored at 12 weeks
The % of completely healed wounds | 12 weeks
Classification of Staphylococcus isolates as MSSA or MRSA resistant | 4 weeks
  MSSA: Methicillin-susceptible Staphylococcus aureus MRSA: Methicillin-resistant Staphylococcus aureus
  What is reported is a binary result: isolates are classified as either "MSSA" or "MRSA"
Classification of Staphylococcus isolates as MSSA or MRSA resistant | at modification of the first-line treatment or new antibiotic prescription (if any; most likey at 14 days and before 12 weeks)
  MSSA: Methicillin-susceptible Staphylococcus aureus MRSA: Methicillin-resistant Staphylococcus aureus
  What is reported is a binary result: isolates are classified as either "MSSA" or "MRSA"
Classification of Staphylococcus isolates as MSSA or MRSA resistant | at week 12 if the wound is still not healed
  MSSA: Methicillin-susceptible Staphylococcus aureus MRSA: Methicillin-resistant Staphylococcus aureus
  What is reported is a binary result: isolates are classified as either "MSSA" or "MRSA"
Classification of Staphylococcus isolates according to clonal complexes (virulence classification) | 4 weeks
Classification of Staphylococcus isolates according to clonal complexes (virulence classification) | at modification of the first-line treatment or new antibiotic prescription (if any; most likey at 14 days and before 12 weeks)
Classification of Staphylococcus isolates according to clonal complexes (virulence classification) | at week 12 if the wound is still not healed
Presence/absence of non-Staphylococcus aureus bacteria that are antibiotic-resistant | week 0
Presence/absence of non-Staphylococcus aureus bacteria that are antibiotic-resistant | week 4
Presence/absence of non-Staphylococcus aureus bacteria that are antibiotic-resistant | at modification of the first-line treatment or new antibiotic prescription (if any; most likey at 14 days and before 12 weeks)
Presence/absence of non-Staphylococcus aureus bacteria that are antibiotic-resistant | at week 12 if the wound is still not healed
Wound microbiota: OTU richness | week 0
  OTU: Operational Taxonomic Unit
Wound microbiota: OTU richness | week 4
  OTU: Operational Taxonomic Unit
Wound microbiota: OTU richness | at modification of the first-line treatment or new antibiotic prescription (if any; most likey at 14 days and before 12 weeks)
  OTU: Operational Taxonomic Unit
Wound microbiota: OTU richness | at week 12 if the wound is still not healed
  OTU: Operational Taxonomic Unit
Wound microbiota: Shannon's Diversity | week 0
Wound microbiota: Shannon's Diversity | week 4
Wound microbiota: Shannon's Diversity | at modification of the first-line treatment or new antibiotic prescription (if any; most likey at 14 days and before 12 weeks)
Wound microbiota: Shannon's Diversity | at week 12 if the wound is still not healed
Wound microbiota: Functional richness | week 0
Wound microbiota: Functional richness | week 4
Wound microbiota: Functional richness | at modification of the first-line treatment or new antibiotic prescription (if any; most likey at 14 days and before 12 weeks)
Wound microbiota: Functional richness | at week 12 if the wound is still not healed
Wound microbiota: Functional diversity | week 0
Wound microbiota: Functional diversity | week 4
Wound microbiota: Functional diversity | at modification of the first-line treatment or new antibiotic prescription (if any; most likey at 14 days and before 12 weeks)
Wound microbiota: Functional diversity | at week 12 if the wound is still not healed
Wound microbiota: the relative abundance of Staphylococcus relative to other bacteria in the wound | week 0
Wound microbiota: the relative abundance of Staphylococcus relative to other bacteria in the wound | week 4
Wound microbiota: the relative abundance of Staphylococcus relative to other bacteria in the wound | at modification of the first-line treatment or new antibiotic prescription (if any; most likey at 14 days and before 12 weeks)
Wound microbiota: the relative abundance of Staphylococcus relative to other bacteria in the wound | at week 12 if the wound is still not healed
Wound microbiota: the number of Staphylococcus strains in a wound | week 0
Wound microbiota: the number of Staphylococcus strains in a wound | week 4
Wound microbiota: the number of Staphylococcus strains in a wound | at modification of the first-line treatment or new antibiotic prescription (if any; most likey at 14 days and before 12 weeks)
Wound microbiota: the number of Staphylococcus strains in a wound | at week 12 if the wound is still not healed
Wound microbiota: the relative abundance of Staphylococcus aureus relative to other bacteria in the wound | week 0
Wound microbiota: the relative abundance of Staphylococcus aureus relative to other bacteria in the wound | week 4
Wound microbiota: the relative abundance of Staphylococcus aureus relative to other bacteria in the wound | at modification of the first-line treatment or new antibiotic prescription (if any; most likey at 14 days and before 12 weeks)
Wound microbiota: the relative abundance of Staphylococcus aureus relative to other bacteria in the wound | at week 12 if the wound is still not healed
Wound microbiota: the relative abundance of Staphylococcus aureus relative to other Staphylococcus in the wound | week 0
Wound microbiota: the relative abundance of Staphylococcus aureus relative to other Staphylococcus in the wound | week 4
Wound microbiota: the relative abundance of Staphylococcus aureus relative to other Staphylococcus in the wound | at modification of the first-line treatment or new antibiotic prescription (if any; most likey at 14 days and before 12 weeks)
Wound microbiota: the relative abundance of Staphylococcus aureus relative to other Staphylococcus in the wound | at week 12 if the wound is still not healed
Wound microbiota: ordination scores on each of two principal components extracted from UniFrac distances between all bacterial samples taken during the study | week 0
Wound microbiota: ordination scores on each of two principal components extracted from UniFrac distances between all bacterial samples taken during the study | week 4
Wound microbiota: ordination scores on each of two principal components extracted from UniFrac distances between all bacterial samples taken during the study | at modification of the first-line treatment or new antibiotic prescription (if any; most likey at 14 days and before 12 weeks)
Wound microbiota: ordination scores on each of two principal components extracted from UniFrac distances between all bacterial samples taken during the study | at week 12 if the wound is still not healed
The presence/absence of anti-phage antibodies in plasma samples | week 0
The presence/absence of anti-phage antibodies in plasma samples | week 4
The presence/absence of anti-phage antibodies in plasma samples | at modification of the first-line treatment or new antibiotic prescription (if any; most likey at 14 days and before 12 weeks)
The presence/absence of anti-phage antibodies in plasma samples | at week 12 if the wound is still not healed

CONTACTS AND LOCATIONS:
Overall Officials: Albert Sotto, MD, PhD, Study Director — Centre Hospitalier Universitaire de Nîmes
Locations (9):
- France (9):
  - CHU de Bordeaux - Hôpital Pellegrin, Bordeaux
  - CHRU de Nîmes - Hôpital Universitaire de Réadaptation du Grau du Roi, Le Grau-du-Roi
  - CHU de Nantes - Hôtel Dieu, Nantes
  - APHP - Hôpital Lariboisière, Paris
  - APHP - Groupe Hospitalier Pitié-Salpetrière, Paris
  - CHRU de Toulouse - Hôpital de Rangueil, Toulouse
  - CH de Tourcoing, Tourcoing
  - Institut Robert Merle d'Aubigné, Valenton
  - CH Intercommunal de Villeneuve-Saint-Georges, Villeneuve-Saint-Georges